CLINICAL TRIAL: NCT02378129
Title: Evaluation of the Effectiveness of Dentin Hypersensitivity Treatment Using Glass Ionomer Cements: A Randomized Clinical Trial
Brief Title: Evaluation of Dentin Hypersensitivity Using Glass Ionomer Cements
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Rafael Guerra Lund, Associate Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPel
Record Dates: First submitted 2015-02-22; First posted 2015-03-04 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin Sensitivity; Dentin Desensitizing Agents; Glass Ionomer Cements; Randomized Controlled Trial
MeSH Terms: conditions — Dentin Sensitivity | interventions — Vidrion-R

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinpro XT (3M ESPE, Minnesota, USA) (Experimental): Resin-modified glass ionomer cement
  Interventions: Drug: Resin-modified glass ionomer cement Clinpro XT
- Vidrion R (SS White, Gloucester, UK) (Active Comparator): Conventional glass ionomer cement
  Interventions: Drug: Glass Ionomer cement Vidrion R

INTERVENTIONS:
Drug: Resin-modified glass ionomer cement Clinpro XT — Clinpro XT (3M ESPE, Minnesota, USA)
  Other Names: Clinpro XT (3M Espe, USA)
  Arms: Clinpro XT (3M ESPE, Minnesota, USA)
Drug: Glass Ionomer cement Vidrion R — Vidrion R (SS White, Gloucester, UK)
  Other Names: Vidrion R (SS White, Gloucester, UK)
  Arms: Vidrion R (SS White, Gloucester, UK)

SUMMARY:
The aim of this randomized, double-blind, split-mouth clinical trial is to evaluate and compare the desensitizing efficacies of the resin-modified glass ionomer cement ClinproTM XT (3M ESPE, Minnesota, USA) and the conventional glass ionomer cement Vidrion R (SS White, Gloucester, UK) at 2-year follow-up.

DETAILED DESCRIPTION:
Subjects will require to have at least two teeth in different hemiarchs with dentin hypersensitivity. Teeth will be randomized into 2 groups, receiving either Clinpro XT or the conventional glass ionomer cement Vidrion R. Prior to the desensitizing treatment (baseline), painful symptoms will be assessed by tactile and air blast tests using the Visual Analogue Scale (VAS). Treatment evaluations will be conducted up to 2-year post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 70 years old
* At least 2 teeth with dentin hypersensitivity in two different hemiarchs
* Dental elements with hypersensitivity without any pulp alteration
* People who are not taking any medication and women who are not pregnant
* Patients without eating disorders or very acidic diets.

Exclusion Criteria:

* Teeth with hypersensitivity that presented extensive or unsatisfactory restorations, fractures, periodontal alterations, caries lesions, orthodontic brackets, endodontic treatments, pulp alterations.
* Subjects who received any desensitizing therapy during the last 3 months
* Subjects being under analgesics/anti-inflammatory drugs at the time of the study
* Teeth with hypersensitivity and non-carious cervical lesions

Ages: 28 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Pain Scores as measured by the Visual Analog Scale (VAS) | Change from Baseline in Pain Scores at 20 minutes; at 7, 15, 21, 30 days; and after 3, 6, 12, 24 months.
  Tactile and air blast tests to evaluate pain with VAS

CONTACTS AND LOCATIONS:
Overall Officials: Rafael G Lund, PhD, Principal Investigator — Federal University of Pelotas

IPD SHARING:
Plan to Share IPD: No
After completing the study, the 20 volunteers continued to be served sporadically at the regular dentistry service of the Faculty of Dentistry of Pelotas, Federal University of Pelotas (UFPel).

REFERENCES:
- [Background] Lund RG, Silva AF, Piva E, Da Rosa WL, Heckmann SS, Demarco FF. Clinical evaluation of two desensitizing treatments in southern Brazil: A 3-month follow-up. Acta Odontol Scand. 2013 Nov;71(6):1469-74. doi: 10.3109/00016357.2013.770919. Epub 2013 Jul 3. PMID 24180588
- [Background] Brannstrom M. The hydrodynamics of the dental tubule and pulp fluid: its significance in relation to dentinal sensitivity. Annu Meet Am Inst Oral Biol. 1966;23:219. No abstract available. PMID 5228880
- [Background] da Rosa WL, Lund RG, Piva E, da Silva AF. The effectiveness of current dentin desensitizing agents used to treat dental hypersensitivity: a systematic review. Quintessence Int. 2013 Jul;44(7):535-46. doi: 10.3290/j.qi.a29610. PMID 23616976
- [Background] Que K, Guo B, Jia Z, Chen Z, Yang J, Gao P. A cross-sectional study: non-carious cervical lesions, cervical dentine hypersensitivity and related risk factors. J Oral Rehabil. 2013 Jan;40(1):24-32. doi: 10.1111/j.1365-2842.2012.02342.x. Epub 2012 Aug 7. PMID 22882712
- [Background] Orchardson R, Gillam DG. Managing dentin hypersensitivity. J Am Dent Assoc. 2006 Jul;137(7):990-8; quiz 1028-9. doi: 10.14219/jada.archive.2006.0321. PMID 16803826
- [Background] Madruga MM, Silva AF, Rosa WL, Piva E, Lund RG. Evaluation of dentin hypersensitivity treatment with glass ionomer cements: A randomized clinical trial. Braz Oral Res. 2017 Jan 5;31:e3. doi: 10.1590/1807-3107BOR-2017.vol31.0003. PMID 28076496